CLINICAL TRIAL: NCT01148602
Title: The CLOQS Trial - Countdown Lights to Optimize Quality in Stroke
Acronym: CLOQS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other); Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Dr. Richard H. Swartz, Dr., Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: UTSP Innovation
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Acute Stroke
Keywords: Acute stroke; Emergency departments; Quality Improvement; Improved Processes; tPA; door-to-needle; door-to-treatment
MeSH Terms: conditions — Stroke; Emergencies | interventions — E1A-Associated p300 Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 'Off Clock' (No Intervention): Stopwatch timers will NOT be used for "off clock" weeks, so patients presenting with hyperacute stroke will be managed normally without the visual timer.
- 'On Clock" (Active Comparator): LED stopwatch-clock timers will be posted for all patients presenting during "ON clock" weeks. All patients presenting with hyperacute stroke will be managed normally with the addition of a visual stopwatch timer.
  Interventions: Other: LED stopwatch-clock timers

INTERVENTIONS:
Other: LED stopwatch-clock timers — We will attach a large, "in-your-face" red LED stopwatch-clock timers to the patient's stretcher at the moment of ED arrival to act as a constant visual reminder to all team members (physicians, RN's, CT technologists) of the urgency of the situation.
  Other Names: Clocks; CLOQS; Clock; LED countdown timer
  Arms: 'On Clock"

SUMMARY:
To reduce door-to-needle times in acute stroke treatment. Using an organizational behaviour intervention (a large stopwatch), we will post a visual cue to remind all parties that "time is brain". We hypothesize that this simple visual cue will improve door-to-CT scan times and door-to-needle treatment times, and thus improve treatment response, and reduce adverse events.

DETAILED DESCRIPTION:
We will construct a large, "in-your-face" red LED stopwatch-clock that is the intervention. The clock will be attached to the stretcher of patients presenting for hyperacute stroke treatment (consideration of tissue plasminogen activator (tPA) treatment at the moment of their Emergency department arrival. This will act as a constant visual reminder to all team members (physicians, RN's, CT technologists) of the urgency of the situation. The study will be a block randomization, by week of presentation. All patients presenting during "on" weeks will have a stopwatch timer with them during the hyperacute stroke workup. During "off" weeks, the clocks will not be used.

ELIGIBILITY:
Inclusion Criteria:

* All patients who present to the emergency room with acute stroke for consideration of treatment with tPA.

Exclusion Criteria:

* Patients presenting to the emergency room (door time) more than 4.5 hours after symptom onset

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3452 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Improved door-to-CT and door-to-needle times. | 18 months
  Improved door-to-CT scan times and door-to-needle treatment times with tPA, with potentially improved response to treatment and reduction in adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Swartz, MD, Principal Investigator — University of Toronto Stroke Program
Locations (3):
- Canada (3):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - University Health Network - Toronto Western Hospital, Toronto, Ontario